CLINICAL TRIAL: NCT02730117
Title: Does Early Initiation of Renal Replacement Therapy Have an Impact on 7-day Fluid Balance in Critically Ill Patients With Acute Kidney Injury With Positive Furosemide Stress Test?: a Multicenter Randomized Controlled Trial
Brief Title: Furosemide Stress Test Guiding Initiation of Renal Replacement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Director of Excellence Center for Critical Care Nephrology, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB.006/59
Record Dates: First submitted 2016-03-18; First posted 2016-04-06 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Furosemide stress test; critical care
MeSH Terms: conditions — Acute Kidney Injury | interventions — Dialysis; Continuous Renal Replacement Therapy; Ventilators, Mechanical; Anti-Bacterial Agents; Cephalosporins; Carbapenems; Vasoconstrictor Agents; Norepinephrine; Dopamine; Milrinone; Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early renal replacement therapy (Experimental): Dialysis with continuous renal replacement therapy machine e.g. Aquarius, Prismaflex, Infomed, starting within 12 hours after randomization
  Patients will receive standard treatments such as anti-bacterial agents, mechanical ventilator, vasopressors as appropriate
  Interventions: Device: Dialysis with continuous renal replacement therapy; Device: Mechanical ventilator; Drug: Anti-Bacterial Agents; Drug: Vasopressors
- Conventional renal replacement therapy (Placebo Comparator): Dialysis with continuous renal replacement therapy machine e.g. Aquarius, Prismaflex, Infomed, after the patients reached at least one of the following criteria;
  1. pH < 7.15 or serum HCO3 < 15 mEq/L
  2. serum K >= 6 mEq/L
  3. Signs of volume overload or P/F ratio < 200
  4. BUN > 60 mg/dL
  Patients will receive standard treatments such as anti-bacterial agents, mechanical ventilator, vasopressors as appropriate
  Interventions: Device: Dialysis with continuous renal replacement therapy; Device: Mechanical ventilator; Drug: Anti-Bacterial Agents; Drug: Vasopressors

INTERVENTIONS:
Device: Dialysis with continuous renal replacement therapy — Continuous renal replacement therapy is a form of 24-hour dialysis in the ICU
Device: Mechanical ventilator — Invasive or noninvasive form of respiratory support
Drug: Anti-Bacterial Agents — Antibacterial agents deemed appropriate by physicians in the ICU
  Other Names: cephalosporin; carbapenem
Drug: Vasopressors — Vasopressors such as Norepinephrine, dopamine, milrinone, dobutamine
  Other Names: Norepinephrine; Dopamine; Milrinone; Dobutamine

SUMMARY:
Does Early Initiation of Renal Replacement Therapy Have an Impact on 7-day Fluid Balance in Critically Ill Patients with Acute Kidney Injury with Positive Furosemide Stress Test?: a Multicenter Randomized Controlled Trial

DETAILED DESCRIPTION:
The objective is to determine if early initiation of renal replacement therapy guided by positive furosemide stress test has an impact on 7-day fluid balance in critically ill patients with acute kidney injury

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years old and admission in an ICU
* Acute kidney injury (defined by serum creatinine increase ≥ 0.3 mg/dL or urine output ≤ 0.5 mL/kg/hour according to KDIGO criteria)
* Informed consent provided by the patient or person with decisional responsibility
* Indwelling bladder catheter
* Documented cause of acute kidney injury from acute tubular necrosis e.g. presence of granular or epithelial casts on urine sediment, FeNa more than 1%, Feurea more than 50%, urine or plasma neutrophil gelatinase-associated lipocalin (NGAL) more than 150 mg/dL
* Opinion of the treating clinical team that patient was well resuscitated and sufficiently clinically stable for the intervention or by noninvasive or invasive measurements i.e. fluid accumulation at least 5% plus at least one of the following e.g. chest radiography, central venous pressure ≥ 8 mmHg, pulse pressure variation < 13%, inferior vena cava collapsibility index < 50% in spontaneously breathing patients or distensibility index < 18% in mechanically ventilated patients

Exclusion Criteria:

* Baseline serum creatinine ≥ 2 mg/dL (male) and ≥ 1.5 mg/dL (female) within 3 months
* Evidence of volume depletion at the time of furosemide administration or active bleeding
* Evidence of obstructive uropathy, renal vein thrombosis or renal artery stenosis, thrombotic microangiopathy, glomerulonephritis, tumor lysis syndrome
* History of renal allograft
* Known pregnancy
* Allergy or known sensitivity to loop diuretics
* Need for emergency renal replacement therapy at randomization or evaluation by the clinical team that the renal replacement therapy should be deferred
* Patient is moribund with expected death within 24 hr or whom survival to 28 days is unlikely due to an uncontrollable comorbidity (cardiac, pulmonary or hepatic end-stage disease; hepatorenal syndrome; poorly controlled cancer; severe post-anoxic encephalopathy; etc.)
* Patients with advance directives issued expressing the desire not to be resuscitated
* Prior treatment with RRT within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Renal replacement therapy proportion | 28 days
  Proportion of patients with FST responsiveness and nonresponsiveness who had received RRT

SECONDARY OUTCOMES:
28-day mortality measured by number of deceased patients at 28-day after the enrollment | 28-day or until hospital discharge
  28-day mortality measured by number of deceased patients at 28-day after the enrollment
ICU-free days measured by number of days (28 days minus ICU length of stay) | through study completion, an average of 28 days
  28 days minus by ICU length of stay
mechanical ventilator-free days measured by number of days (28 days minus days using mechanical ventilator) | through study completion, an average of 28 days
  28 days minus by days using mechanical ventilator
dialysis dependence measured by need for renal replacement therapy in 28 days | through study completion, an average of 28 days
  dialysis dependence at hospital discharge
7-day fluid balance | 7 days
  7-day fluid balance
RRT free days | through study completion, an average of 28 days
  28 days minus by days on RRT
Length of ICU stay | through study completion, an average of 28 days
  Length of ICU stay
Length of hospital stay | through study completion, an average of 28 days
  Length of hospital stay
Renal recovery | through study completion, an average of 28 days
  Urine output > 1,000 ml without diuretics or > 2,000 ml with diuretics
Adverse events | through study completion, an average of 28 days
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nattachai Srisawat, MD, Principal Investigator — Excellence Center of Critical Care Nephrology, Chulalongkorn University
Locations (1):
- Sasipha Tachaboon, Bangkok, Pathumwan, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Lumlertgul N, Peerapornratana S, Trakarnvanich T, Pongsittisak W, Surasit K, Chuasuwan A, Tankee P, Tiranathanagul K, Praditpornsilpa K, Tungsanga K, Eiam-Ong S, Kellum JA, Srisawat N; FST Study Group. Early versus standard initiation of renal replacement therapy in furosemide stress test non-responsive acute kidney injury patients (the FST trial). Crit Care. 2018 Apr 19;22(1):101. doi: 10.1186/s13054-018-2021-1. PMID 29673370